CLINICAL TRIAL: NCT00753012
Title: An In Depth Cardiovascular Study of Lisdexamfetamine (LDX; Vyvanse) in Healthy and Treated Hypertensive Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Cardiovascular Study of Lisdexamfetamine in Healthy and Hypertensive Attention Deficit Hyperactivity Disorder Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Paul Hammerness, MD, Assistant Professor Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2008-P-000121
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Results first posted 2012-09-24 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-08

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: cardiovascular testing; home blood pressure monitoring; office home blood pressure monitoring; cardiopulmonary exercise testing; transthoracic echocardiography; Lisdexamfetamine; Vyvanse; normotensive and hypertensive adults with ADHD; ADHD medication.
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lisdexamfetamine (Experimental): Adults who meet DSM-IV-TR criteria for ADHD.
  Group 1 is normotensive adults; Group 1 does not have high blood pressure. Group 2 is primary hypertensive adults; Group 2 does have high blood pressure and is being treated with stable doses of hypertensive medications achieving a blood pressure of <135/85.
  Interventions: Drug: Lisdexamfetamine

INTERVENTIONS:
Drug: Lisdexamfetamine — Lisdexamfetamine daily until the completion of participation in the clinical trial (up to Week 11 or final study visit). Subjects will start on 30 mg of LDX per day for the first week of treatment. The dose will be increased weekly in 20 mg increments, up to a 70 mg daily (maximum). If significant adverse effects (AE) occur, the daily dose may be reduced by 20 mg. At subsequent visits, a higher dose may be resumed if tolerated. Both cohorts of the study will follow the same treatment plan.
  Other Names: Vyvanse

SUMMARY:
The purpose of this research study is to learn about the effects of a medication called Vyvanse on the heart (cardiovascular system). The U.S. Food and Drug Administration (FDA) has approved Vyvanse for the treatment of Attention Deficit Hyperactivity Disorder (ADHD). People who have ADHD have trouble paying attention, organizing, and planning; these symptoms can cause problems at work, socially and at home.

Vyvanse (also known as Lisdexamfetamine) is a stimulant class medication. There have been reports of serious cardiovascular effects in children and adults treated with stimulants. While there is no definite evidence that these events were related to the use of stimulants, the deaths have raised questions about the cardiovascular safety of stimulants.

The study will involve in-depth cardiovascular tests, namely echocardiograph (ultrasound of the heart) and cardiopulmonary exercise test (also called stress test; subjects exercise on a bicycle while measuring their heart activity and breathing is monitored by cardiologists).

The investigators predict to see changes in blood pressure and heart rate as shown in previous clinical studies, and that the in-depth cardiovascular tests will provide new insights into the cardiovascular impact of stimulants.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients 18-60 years of age.
2. A current DSM-IV-TR diagnosis of ADHD, confirmed by the Adult ADHD Clinical Diagnostic Scale (ACDS) at Screening.
3. In phase two only; Stage I primary hypertension (SBP 140-159 mm Hg/DBP 90-99 mm Hg) as defined by Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (Chobanian et al, 2003).
4. In phase two only; Treatment with stable doses of up to two FDA approved antihypertensive medications achieving a stable blood pressure of <135/85. Acceptable classes of medications include diuretics, beta-blockers, angiotensin-converting-enzyme (ACE) inhibitors or receptor blockers, aldosterone antagonists, calcium-channel blockers (Rosendorff et al, 2007).

Exclusion Criteria:

1. Pregnant or nursing females.
2. Clinically significant cardiovascular history, including angina, syncope, thrombosis, aneurysm, myocardial infarction, myocarditis, valvular disease, heart failure, or arrhythmia. Hypertension is exclusionary in phase one subjects.
3. In phase two; hypertension is not exclusionary, however blood pressure with antihypertensive treatment of ≥135/85 at baseline is exclusionary.
4. Clinically significant or unstable medical condition including pulmonary (asthma, edema, thrombosis), renal, hepatic, metabolic (thyroid) or neurological disorder, based upon a medical history.
5. Orthopedic impairment or BMI that significantly impacts or restricts exercise performance testing, per clinician judgment.
6. Any clinically unstable psychiatric conditions including suicidality, homicidality, bipolar disorder, psychosis.
7. Current (within 3 months) DSM-IV-TR criteria for current abuse or dependence with any psychoactive substance other than nicotine, including alcohol, prescription medicines and/or street drugs. In addition, subjects with clinically significant histories of dependence on alcohol, prescription medications or "street drugs" will be excluded, if such history places subjects at heightened risk, and/or may be associated with cardiovascular sequelae, based on clinician judgment.
8. Ongoing treatment with any psychotropic medication, including anxiolytics, antidepressants, mood stabilizers.
9. Use of Monoamine Oxidase Inhibitors (MAOIs) including linezolid within two weeks prior to starting study medication.
10. Mental retardation (IQ < 75).
11. History of intolerance or allergy to LDX.
12. Diagnosis of glaucoma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hammerness, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Normotensive Adults With ADHD: Group 1 is comprised of adults who meet DSM-IV-TR criteria for ADHD and do not have high blood pressure.
- Primary Hypertensive Adults With ADHD: Group 2 is comprised of adults who meet the full DSM-IV criteria for ADHD, and who also high blood pressure being treated with stable doses of up to two FDA approved hypertensive medications to achieve a stable blood pressure of <135/85. High blood pressure is defined as 140-159mmHg/90-99 mmHg.
Period: Overall Study
Arm/Group | Normotensive Adults With ADHD | Primary Hypertensive Adults With ADHD
Started | 15 | 9
Completed | 7 | 8
Not Completed | 8 | 1
Not completed — Ineligible, abnormal cardiac histo | 1 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 4 | 0
Not completed — Confounded endpoint data | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normotensive Adults With ADHD | Primary Hypertensive Adults With ADHD | Total
Number analyzed (Participants) | 15 | 9 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 9 | 24
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.80 (11.59) | 51.33 (7.87) | 41.00 (13.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 15 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricle Size
Description: Size of the heart's left ventricle chamber (Left Ventricular End Diastolic Dimension; LVEDD) following 3-6 months of stimulant medication, according to cardiac ultrasound (transthoracic echocardiogram; TTE)
Time Frame: 3-6 months
Population: 14 subjects completed endpoint TTE; one HTN subject missed the scheduled endpoint TTE appointment.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Normotensive Adults With ADHD | Primary Hypertensive Adults With ADHD
Number analyzed (Participants) | 7 | 7
mm | 44.42 (7.07) | 43.57 (6.13)

2. Primary Outcome: Cardiac Function Index (E/A Ratio)
Description: Left ventricle diastolic function index, following 3-6 months of stimulant medication, according to cardiac ultrasound (transthoracic echocardiogram; TTE)
Time Frame: 3-6 months
Measure: Mean (Standard Deviation); unit: cm/sec/cm/sec
Arm/Group | Normotensive Adults With ADHD | Primary Hypertensive Adults With ADHD
Number analyzed (Participants) | 7 | 7
cm/sec/cm/sec | 1.38 (0.48) | 1.36 (0.84)

3. Primary Outcome: Blood Pressure at Maximum Exertion
Description: Diastolic blood pressure (DBP) at maximum exertion following 3-6 months of stimulant medication, according to cardiopulmonary exercise testing (CPET)
Time Frame: 3-6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Normotensive Adults With ADHD | Primary Hypertensive Adults With ADHD
Number analyzed (Participants) | 7 | 8
mmHg | 80.43 (11.97) | 85.00 (8.07)

ADVERSE EVENTS:
Arm/Group | Normotensive Adults With ADHD | Primary Hypertensive Adults With ADHD
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/8
Other Adverse Events (participants affected / at risk) | 11/14 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 4.2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normotensive Adults With ADHD (N=14) | Primary Hypertensive Adults With ADHD (N=8)
anxiety (Psychiatric disorders) | 2 (23) | 3 (39)
back pain (General disorders) | 2 (7) | 0 (0)
blind spot (Eye disorders) | 0 (0) | 1 (14)
blurred vision (Eye disorders) | 1 (3) | 0 (0)
cold symptoms (General disorders) | 5 (18) | 1 (7)
congestion (Respiratory, thoracic and mediastinal disorders) | 4 (12) | 1 (16)
constipation (Gastrointestinal disorders) | 1 (23) | 1 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6)
depressed mood (Psychiatric disorders) | 1 (1) | 1 (30)
difficulty achieving erection (Reproductive system and breast disorders) | 1 (43) | 0 (0)
dry mouth (General disorders) | 6 (78) | 4 (164)
dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (7)
feelings of self-consciousness (Psychiatric disorders) | 1 (7) | 0 (0)
fever (General disorders) | 0 (0) | 1 (12)
feeling flustered (Psychiatric disorders) | 0 (0) | 1 (7)
foot pain (General disorders) | 0 (0) | 1 (11)
GI upset (Gastrointestinal disorders) | 1 (1) | 0 (0) — Gastrointestinal upset
hand tremor (General disorders) | 1 (3) | 0 (0)
headache (General disorders) | 8 (22) | 2 (6)
heartburn (General disorders) | 1 (3) | 2 (6)
increased energy (General disorders) | 1 (5) | 2 (60)
insomnia (General disorders) | 3 (8) | 6 (19)
irritability (Psychiatric disorders) | 2 (11) | 1 (1)
jaw tension (General disorders) | 2 (18) | 2 (132)
jittery (General disorders) | 5 (27) | 1 (14)
lightheadedness (General disorders) | 1 (2) | 1 (2)
lip swelling (General disorders) | 0 (0) | 1 (2)
low appetite (Metabolism and nutrition disorders) | 5 (111) | 1 (2)
low energy (General disorders) | 2 (5) | 0 (0)
muscle aches (Musculoskeletal and connective tissue disorders) | 3 (70) | 0 (0)
muscle tension (Musculoskeletal and connective tissue disorders) | 2 (21) | 0 (0)
muscle twitch (Musculoskeletal and connective tissue disorders) | 2 (7) | 0 (0)
nausea (General disorders) | 0 (0) | 3 (11)
numbness (General disorders) | 0 (0) | 1 (1)
racing (General disorders) | 1 (14) | 2 (5) — Feeling 'on the go' or 'driven by a motor'
sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (7)
tension (General disorders) | 0 (0) | 1 (3)
tightness in the hand (General disorders) | 1 (1) | 0 (0)
urinary tract infection (Renal and urinary disorders) | 1 (2) | 0 (0)
viral illness (Infections and infestations) | 1 (14) | 0 (0)
vomiting (Gastrointestinal disorders) | 2 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No